CLINICAL TRIAL: NCT05749705
Title: Fat to Lean Mass Ratio and Its Effect on Low Back Pain and Permanent Functional Disability.
Status: Completed | Type: Observational
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, Mohamed Moustafa Mohamed Ahmed, Assistant Professor, University of Jazan
Other Study IDs: 94177
Record Dates: First submitted 2023-02-18; First posted 2023-03-01 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Low Back Pain, Mechanical
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Fat to Lean Mass Ratio — The study will be conducted for people who suffer from excess fat mass and their age is over 18 years.
  years will be calculated with G power

SUMMARY:
The study was conducted for people who suffer from excess fat mass and their age is over 18 years will be calculated with G*power will be used body composition analyzer to calculate the percentage of fat.

DETAILED DESCRIPTION:
Cross-sectional study was applied. Data was collected through a questionnaire (oswestry disability index arabic version). Fat percentage was taken by Body composition analyzer.

ELIGIBILITY:
Inclusion Criteria:

* Excess fat mass
* Age must be over 18 years.

Exclusion Criteria:

* People under the age of 18.
* Low back pain not associated with increased fat mass.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: People who suffer from excess fat mass and their age is over 18 years.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2023-02-05 (Actual); Primary Completion 2023-03-05 (Actual); Study Completion 2023-03-12 (Actual)

PRIMARY OUTCOMES:
Fat to Lean mass ratio | Immediately after the admission
  Body composition analyzer will be used to measure the percentage of fat

SECONDARY OUTCOMES:
Low Back Pain and disability | Immediately after the admission
  Oswestry disability index arabic version will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Jazan University, Jizan, Gizan, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No